CLINICAL TRIAL: NCT06617637
Title: Comparison of the Effects of Aerobic-Based Virtual Reality Exercise Training (Exergame) and Traditional Aerobic Exercise Training on Physical Fitness, Functional Capacity and Cognitive Function in Individuals with Down Syndrome: (DOWNFIT)
Brief Title: Effects of Aerobic-Based Virtual Reality Exercise Training and Traditional Aerobic Exercise Training on Physical Fitness, Functional Capacity and Cognitive Function in Individuals with Down Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Alis Kostanoğlu Asoc.Prof., Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24/09/2024 - BezmialemVU
Record Dates: First submitted 2024-09-24; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Down Syndrome; Aerobic Exercise; Virtual Reality Based Therapy; Exergame; Physical Fitness; Functional Capacity; Cognitive Function
Keywords: Down Syndrome; Aerobic exercise; Virtual reality; Exergame; Physical Fitness; Functional Capacity; Cognitive function
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Participants to be included in the study will be randomly grouped into three groups. Two groups will be the intervention group and one group will be the control group.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers conducting the evaluations in the study will be masked to the treatment groups, and the researcher conducting the statistical analysis will be masked to the evaluations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic-Based Virtual Reality Exercise Training Group (Experimental): Aerobic exercise training will be applied to the aerobic-based virtual reality exercise group with an Xbox Kinect 360 (Microsoft, Washington, USA) for 20 sessions, 2 days a week, for 10 weeks.
  Interventions: Other: Aerobic Based Virtual Reality Exercise Training
- Traditional Aerobic Exercise Training Group (Active Comparator): The traditional aerobic exercise group will receive treadmill training under the supervision of a physiotherapist 2 days a week for 10 weeks.
  Interventions: Other: Traditional Aerobic Exercise Training
- Control Group (No Intervention): Participants in the control group will be advised to continue with their standard daily living activities.

INTERVENTIONS:
Other: Aerobic Based Virtual Reality Exercise Training — With Aerobic Based Virtual Reality Exercise Training, participants will perform aerobic exercise training with the Xbox Kinect 360 game "Your Shape Fitness Evolved 2012". "Your Shape Fitness Evolved 2012" is a game that requires basic coordination and is designed to improve the fitness levels of individuals. The game is used as an entertaining aerobic training tool that includes many aerobic activities such as boxing, yoga, dancing, etc. with adjustable difficulty levels.
  Arms: Aerobic-Based Virtual Reality Exercise Training Group
Other: Traditional Aerobic Exercise Training — Using a treadmill, participants will be put through an exercise training consisting of a 10-minute warm-up at 0 degree incline, a 20-30-minute (by increasing the walking time by 5 minutes at the end of the first four weeks and the beginning of the last four weeks) walking at 40-80% of the heart rate reserve (moderate-vigorous intensity) and a 10-minute cool-down period. Treadmill walking levels will be changed if necessary to ensure the targeted exercise intensity.
  Arms: Traditional Aerobic Exercise Training Group

SUMMARY:
This study aims to investigate the effectiveness of aerobic-based virtual reality exercise training and traditional aerobic exercise training on physical fitness, functional capacity, cognitive functions and quality of life in individuals with Down syndrome.

DETAILED DESCRIPTION:
The most common chromosomal disorder caused by the presence of an extra copy of chromosome 21, resulting in Down syndrome. Individuals with Down syndrome have a higher prevalence of musculoskeletal, neurological, and cardiovascular system problems compared to healthy individuals. Physical activity and exercise play a significant role in the treatment of Down syndrome. Among the preferred exercise programs in treatment, aerobic exercise improves cardiorespiratory functions, has positive effects on physical fitness parameters, enhances quality of life, and improves cognitive function. In addition to traditional aerobic exercise training using devices such as bicycles and treadmills, virtual reality-based aerobic exercise training is also a widely used method. However, there is a lack of studies on the use of aerobic-based virtual reality exercises in individuals with Down syndrome in the literature. The studies available in the literature mainly focus on balance and postural control in virtual reality exercises.

This study aims to investigate the effectiveness of aerobic-based virtual reality exercise training compared to traditional aerobic exercise training on physical fitness, functional capacity, cognitive function, and quality of life in individuals with Down syndrome.

The study plans to include 40 participants with Down syndrome aged between 13 and 18 years. The participants will be divided into three groups: Aerobic-Based Virtual Reality Exercise Training Group, Traditional Aerobic Exercise Training Group and Control Group. The Aerobic-Based Virtual Reality Exercise Training Group will perform aerobic exercise training using Xbox Kinect 360 device, while the Traditional Aerobic Exercise Training Group will use a treadmill for aerobic exercise training. During the exercise training, participants heart rate and oxygen saturation will be monitored using a pulse oximeter, and the training will be supervised by a physiotherapist. The exercise program will be conducted twice a week for a total of 10 weeks. The individuals in the Control Group will be advised to continue their standard daily activities.

The physical fitness components of all participants will be evaluated using the Eurofit Test Battery. The Timed Up and Go Test and 6-Minute Walk Test will be used to assess participants submaximal functional capacities.The Childrens Quality of Life Scale will be used to assess quality of life, and The Behavior Rating Inventory of Executive Function will be used to evaluate cognitive function. To assess physical activity levels and monitor them, the participants will be administered the Godin Leisure-Time Exercise Questionnaire on a weekly basis for 10 weeks. The enjoyment of physical activities by the participants will be evaluated using the Physical Activity Enjoyment Scale.

ELIGIBILITY:
Inclusion Criteria:

* According to DSM-V (Diagnostic and Statistical Manual of Mental Disorders-V) criteria, individuals with Down syndrome with mild to moderate intellectual disability
* Being able to understand the instructions in the assessment and exercise program
* Being willing to participate in the study

Exclusion Criteria:

* Having participated in any structured exercise program in the last 6 months before participating in the study
* Having any heart disease or other chronic physical, behavioral or cognitive problems that limit their participation in the exercise program
* Having severe visual or auditory problems
* Having any history of surgery affecting musculoskeletal structures

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Eurofit Fitness Test Battery | 3 months
  The Eurofit Fitness Test Battery is an assessment method consisting of a series of tests developed by the European Council in the 1980s to assess physical fitness. The Eurofit Test Battery is designed to be performed with simple equipment and in a short time, usually 25-40 minutes. This test battery evaluates different physical fitness components such as balance, speed, flexibility, explosive power, muscular strength, muscular endurance, agility and aerobic endurance. These physical fitness components included in the test are evaluated with different tests.
6-minute Walk Test | 3 months
  The 6-Minute Walk Test (6-MWT) will be used to assess the submaximal functional capacity of the participants. The aim of the 6-Minute Walk Test is to walk the longest distance possible in a 30-meter corridor in 6 minutes. The 6-MWT will be performed in accordance with the guidelines reported by the American Thoracic Society.
Behavioral Rating Inventory Of Executive Function (BRIEF) | 3 months
  The Behavioral Rating Inventory of Executive Function (BRIEF) is a 3-point Likert-type scale with 86 statements indicating specific behaviors. The statements are scored as '1', '2', '3', respectively. A high score indicates a high level of executive dysfunction.

SECONDARY OUTCOMES:
Timed Up and Go Test | 3 months
  The Timed Up and Go Test (TUG) will be used to assess participants' functional capacity, balance and walking speed. In the TUG, the participant is asked to get up from a chair with a seat height of approximately 46 cm, walk 3 meters, turn around and sit back down in the chair. The time it takes the patient to complete this activity gives the result of the test.
Anthropometric Measurement - Body Mass Index | 3 months
  For anthropometric measurement, participants; weight (in kilograms) and height (in meters) will be measured and recorded to calculate body mass index (kg/m^2).
Anthropometric Skinfold Measurement | 3 months
  Total body fat ratio will be obtained by measuring the skin fold in the triceps and subscapular anatomical regions with a special caliper called skinfold. To determine the visceral fat ratio, participants waist and hip circumferences will be measured and recorded.
The Pediatric Quality of Life Inventory | 3 months
  The Pediatric Quality of Life Inventory has child and parent forms, each consisting of 23 items, and each item is scored between 0-100. The child/adolescent is asked to mark the most appropriate option for each sentence, and the parent is asked to mark the most appropriate option for their child. A five-choice Likert-type response scale is used throughout the scale. The higher the total score from the scale, the higher the quality of life.
Godin Leisure-Time Exercise Questionnaire | 3 months
  Godin Leisure-Time Exercise Questionnaire will be administered to participants weekly for 10 weeks to assess and monitor their physical activity levels. In this assessment, a score of 24 and above will be classified as "active", a score between 14 and 23 will be classified as "moderately active", and a score of 13 and below will be classified as "not sufficiently active".
Physical Activity Enjoyment Scale | 3 months
  Physical Activity Enjoyment Scale will be used to assess positive emotions such as pleasure and enjoyment expected from physical activities. Participants are asked to indicate the extent to which they agree with each item, using a seven-point scale ranging from 1-strongly disagree to 7-strongly agree. A high average score from the scale indicates a high level of enjoyment from physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: Alis Kostanoğlu, PhD, Principal Investigator — Bezmialem Vakif University; Elif Durgut, PhD, Study Chair — Bezmialem Vakif University; Ayça Arslantürk Yıldırım, MSc, Study Chair — Bezmialem Vakif University; Merve Sevinç Gündüz, MSc, Study Chair — Bezmialem Vakif University; Gökhan Can Törpü, BPT, Study Chair — Bezmialem Vakif University; Abdurrahman Cahit Örengül, PhD, Study Chair — Istanbul University
Locations (1):
- Bezmialem Vakıf University, Istanbul, Eyüpsultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonarakis SE, Skotko BG, Rafii MS, Strydom A, Pape SE, Bianchi DW, Sherman SL, Reeves RH. Down syndrome. Nat Rev Dis Primers. 2020 Feb 6;6(1):9. doi: 10.1038/s41572-019-0143-7. PMID 32029743
- [Background] Shields N. Physiotherapy management of Down syndrome. J Physiother. 2021 Oct;67(4):243-251. doi: 10.1016/j.jphys.2021.08.016. Epub 2021 Sep 10. No abstract available. PMID 34511385
- [Background] Lopes JBP, Duarte NAC, Lazzari RD, Oliveira CS. Virtual reality in the rehabilitation process for individuals with cerebral palsy and Down syndrome: A systematic review. J Bodyw Mov Ther. 2020 Oct;24(4):479-483. doi: 10.1016/j.jbmt.2018.06.006. Epub 2018 Jun 28. PMID 33218550
- [Background] Silva V, Campos C, Sa A, Cavadas M, Pinto J, Simoes P, Machado S, Murillo-Rodriguez E, Barbosa-Rocha N. Wii-based exercise program to improve physical fitness, motor proficiency and functional mobility in adults with Down syndrome. J Intellect Disabil Res. 2017 Aug;61(8):755-765. doi: 10.1111/jir.12384. Epub 2017 Jun 6. PMID 28585394
- [Background] Gomez Alvarez N, Venegas Mortecinos A, Zapata Rodriguez V, Lopez Fontanilla M, Maudier Vasquez M, Pavez-Adasme G, Hemandez-Mosqueira C. [Effect of an intervention based on virtual reality on motor development and postural control in children with Down Syndrome]. Rev Chil Pediatr. 2018 Dec;89(6):747-752. doi: 10.4067/S0370-41062018005001202. Spanish. PMID 30725064